CLINICAL TRIAL: NCT00676299
Title: An Open-label, Phase I Study to Determine the Safety and Pharmacokinetics of JNJ-26483327, a Multi-targeted Kinase Inhibitor, Administered to Subjects With Advanced Stage and/or Refractory Solid Malignancies
Brief Title: A Safety and Dose-finding Study of JNJ-26483327, a Drug in Development for Cancer, for Patients With Advanced and/or Refractory Solid Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011881
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Protein Kinase Inhibitors; Antineoplastic Protocols; Clinical Trial, Phase 1; Maximum Tolerated Dose; Pharmacokinetics; Advanced Malignancies; Solid Malignancies
Keywords: Advanced Solid Cancers; Refractory Solid Cancers; Protein Kinase Inhibitors; Phase 1 Study; Oral Chemotherapy
MeSH Terms: interventions — JNJ-26483327

INTERVENTIONS:
Drug: JNJ-26483327

SUMMARY:
The purpose of this study is to assess JNJ-26483327 (a drug in development for cancer) for the safety of the drug in patients with advanced solid tumors that have not responded or are no longer responding to available therapies. The absorption, breakdown and elimination of the drug will also be studied.

DETAILED DESCRIPTION:
JNJ-26483327, a multi-targeted reversible kinase inhibitor, is a new drug in development for treatment of cancer. This study will test the safety (the effect on the body) of JNJ-26483327 and the highest dose of JNJ-26483327 that patients with advanced cancer can tolerate will be determined. Antitumor activity of JNJ-26481585 will be evaluated.

JNJ-26483327 will be administered in a continuous regimen (orally twice daily) in 28-day treatment cycles. The dose of JNJ-26483327 will start low and will be increased during the study in groups of 1 to 6 patients. If a patient or a group of patients does not have severe side effects, the next group of patients will get a higher dose. The dose will increase until some patients have severe side effects. The dose will then be decreased to a dose level where severe side effects are observed in less than 1/3 of patients. Once a safe dose level has been determined an additional group of 12-18 patients will be treated. The amount of JNJ-26483327 in the blood will be measured and the effect of the disease will be evaluated in all patients.

Patients will be screened for eligibility within 4 weeks before study treatment is given. The treatment will consist of 28-day treatment cycles in a continuous twice daily dosing regimen.

During Cycle 1, patients are required to stay in the hospital for 2-3 nights and 2 full days. In addition there are 5 daytime visits during Cycles 1 and 2 (combined) that may take up to 6 hours after the morning dose. From Cycle 3 onwards, one hospital visit is required for each cycle of treatment.

Throughout the study, especially during Cycles 1 and 2, patients will undergo frequent blood and urine tests, procedures to assess safety including heart function, and tests to assess the course of the patient's illness. The duration of treatment will depend on adverse effects and whether there is benefit from the treatment. Two weeks after the last dose of the study drug, patients are required to return to the study site for follow-up assessments. Patients will take JNJ-26483327 capsules by mouth twice a day throughout treatment. Patients will be allowed to continue at the same dose level as long as there are no unacceptable side effects, and there is benefit to the patient based on the study doctor's evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of solid malignancy that is advanced or refractory and progressing and for which standard treatments do not exist or are no longer effective
* radiological assessment of disease within 4 weeks of first study drug administration
* overall health status as determined by the Eastern Cooperative Oncology Group (ECOG) < = 2
* life expectancy > 3 months
* adequate gastrointestinal absorption and ability to swallow
* left ventricular ejection fraction (LVEF) > 50% and protocol-defined criteria for laboratory tests.

Exclusion Criteria:

* Cancer has spread to the central nervous system
* chemotherapy, radiotherapy, immunotherapy within 4 weeks before study drug administration or incomplete recovery from preceding surgery or toxicity of prior anticancer therapy (excluding peripheral neuropathy and alopecia)
* history of uncontrolled heart disease as defined in the protocol
* history of pulmonary fibrosis
* acute infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Determine the safety (effects on the body) and the maximum tolerated dose of JNJ-26483327 in patients with cancer. Determine how JNJ-26483327 taken by patients as an oral capsule is absorbed, broken down and eliminated.

SECONDARY OUTCOMES:
Assess the anti-cancer activity of JNJ-26483327 in patients with cancer. Determine how JNJ-26483327 works in patients with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.